CLINICAL TRIAL: NCT02038608
Title: Pathophysiology of Non Motor Signs and Compensatory Mechanisms in Parkinson's Disease: Role of the Serotoninergic and Dopaminergic Lesions Studied by PET
Brief Title: Compensatory Mechanisms in Parkinson Disease (PD)
Acronym: CompensationPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012.722
Record Dates: First submitted 2014-01-13; First posted 2014-01-16 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson; serotonin; dopamine; non motor; progression; PET
MeSH Terms: conditions — Parkinson Disease; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET (Experimental)
  Interventions: Device: PET

INTERVENTIONS:
Device: PET

SUMMARY:
Parkinson's disease is characterized by a large number of non motor, especially neuropsychiatric, signs. Their pathophysiology is complex but the role of dopaminergic and serotoninergic systems dysfunction is suggested by several studies. In addition, the serotoninergic system is involved in the pathophysiology of dyskinesias. Very few studies have analyzed the abnormalities of these two neurotransmission systems at disease onset, in de novo PD patients. Furthermore, the parallel evolution of the degeneration of the dopaminergic and serotoninergic systems with disease progression remains unknown. Thus the present study aims at determining, by using PET and 11C-PE2I and 11C-DASB the respective role of the serotoninergic and dopaminergic systems dysfunction in motor and non motor manifestations in PD, at different evolution stages.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Patients presenting doparesponsive Parkinson's disease
* Patient's age between 40 and 70 years old
* Absence of other neurological or psychiatric disease
* Absence of cognitive decline ( MATTIS > 130)
* For women of childbearing age a pregnancy test and a contraceptive method will be required
* Informed consent sign

Healthy subjects

* subject's age between 40 and 70 years old
* Absence of neurological or psychiatric disease
* Absence of cognitive decline ( MATTIS > 130)
* For women of childbearing age a pregnancy test and a contraceptive method will be required
* Informed consent sign

Exclusion Criteria:

Patients

* patient's age < 40 years old or > 70 years old
* Other neurological or psychiatric disease
* Cognitive decline (MATTIS < 130).
* Having participated to a PET or SPECT study in the last 12 months
* Pregnancy
* Severe concomitant disease

Healthy subjects

* subject's age < 40 years old or > 70 years old
* Neurological or psychiatric disease
* Cognitive decline (MATTIS < 130).
* Having participated to a PET or SPECT study in the last 12 months
* Pregnancy
* Severe concomitant disease

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Respective progression of both dopaminergic and serotoninergic lesions in Parkinson's disease | This will be achieved at the end of the inclusion period, thus 24 to 36 months after study onset (January 2014).
  Dopaminergic lesions will be determined by positron emission tomography (PET) using 11C-PE2I in 3 groups of PD patients (de novo; mid-stage (4-7 years of evolution); late-stage (8-10 years of evolution). Serotoninergic lesions will be assessed by positron emission tomography (PET) using 11C-DASB in the same 3 groups of PD patients. In addition a control group will be included.

SECONDARY OUTCOMES:
Correlations between neuropsychiatric observed in Parkinson's disease at different stages of evolution | These correlations will be determined at the end of the inclusion period, thus 24 to 36 months after study onset (January 2014).
  Dopaminergic lesions will be determined by positron emission tomography (PET) using 11C-PE2I in 3 groups of PD patients (de novo; mid-stage (4-7 years of evolution); late-stage (8-10 years of evolution). Serotoninergic lesions will be assessed by positron emission tomography (PET) using 11C-DASB in the same 3 groups of PD patients. In addition a control group will be included.
  The neuropsychiatric manifestations studied are :
  * hypo and hyperdopaminergic signs : ECMP scale
  * Apathy using LARS scale
  * Anxiety using BAI scale
  * Depression using BDI scale (Beck Depression Inventory)
  * Affective well-being and asthenia using visual analogic scales of Norris
  * MATHYS scale
  * Global cognitive scale : MATTIS
  * Food behavior using TFEQ scale
  * Personality : TCI-R scale
  * Impulsivity by UPPS scale
Role of dopaminergic and serotoninergic lesions in fatigue | This will be determined at the end of the inclusion period, thus 24 to 36 months after study onset (January 2014).
  : Dopaminergic lesions will be determined by positron emission tomography (PET) using 11C-PE2I in 3 groups of PD patients (de novo; mid-stage (4-7 years of evolution); late-stage (8-10 years of evolution). Serotoninergic lesions will be assessed by positron emission tomography (PET) using 11C-DASB in the same 3 groups of PD patients. In addition a control group will be included.
  Fatigue will be assessed using the PDFS-16 scale
Relationship between the severity of dopaminergic and serotoninergic lesions and the quality of life | These correlations will be determined at the end of the inclusion period, thus 24 to 36 months after study onset (January 2014).
  Dopaminergic lesions will be determined by positron emission tomography (PET) using 11C-PE2I in 3 groups of PD patients (de novo; mid-stage (4-7 years of evolution); late-stage (8-10 years of evolution). Serotoninergic lesions will be assessed by positron emission tomography (PET) using 11C-DASB in the same 3 groups of PD patients. In addition a control group will be included.
  Fatigue will be assessed using the PDQ39 (Parkinson's Disease Questionnaire) scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Hopital Neurologique Pierre Wertheimer, Bron, France

REFERENCES:
- [Result] Maillet A, Krack P, Lhommee E, Metereau E, Klinger H, Favre E, Le Bars D, Schmitt E, Bichon A, Pelissier P, Fraix V, Castrioto A, Sgambato-Faure V, Broussolle E, Tremblay L, Thobois S. The prominent role of serotonergic degeneration in apathy, anxiety and depression in de novo Parkinson's disease. Brain. 2016 Sep;139(Pt 9):2486-502. doi: 10.1093/brain/aww162. Epub 2016 Aug 17. PMID 27538418